CLINICAL TRIAL: NCT03784755
Title: A Randomized Phase III Trial of Local Ablative Therapy For Hormone Sensitive Oligometastatic Prostate Cancer [PLATON]
Brief Title: Local Ablative Therapy For Hormone Sensitive Oligometastatic Prostate Cancer
Acronym: PLATON
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR20
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer Metastatic
Keywords: Oligometastatic Hormone
MeSH Terms: interventions — Radiosurgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (standard of care) (Active Comparator): Standard systemic therapy
  + Ablative therapy to untreated prostate primary for patients with low volume metastatic disease burden
  Interventions: Other: Standard of care
- Arm 2 (standard systemic therapy + ablative therapy)) (Experimental): Local Ablative therapy to all sites of disease (including untreated prostate primary)
  + Standard systemic therapy
  Interventions: Radiation: Ablative Radiation Therapy; Other: Standard of care

INTERVENTIONS:
Radiation: Ablative Radiation Therapy — Undergo stereotactic radiotherapy and/or surgery to all sites of disease (oligometastases and primary prostate if previously untreated).
  Other Names: SBRT; Stereotactic External Beam Irradiation; Stereotactic Radiation Therapy; Stereotactic Radiotherapy
  Arms: Arm 2 (standard systemic therapy + ablative therapy))
Other: Standard of care — Patients continue to receive their current planned systemic therapy at the discretion of the treating physician

SUMMARY:
The purpose of this study is to compare the effects of ablative therapy (radiation or surgery) to all sites of disease combined with standard treatments on prostate cancer, compared to the standard or usual treatments used to treat this disease.

DETAILED DESCRIPTION:
The standard or usual treatment for this disease is systemic therapy, which includes androgen deprivation therapy (ADT) with or without chemotherapy or hormone therapy. Additionally, for some patients with specific disease features, standard treatment may also include ablative treatment (radiation or surgery) of the prostate gland if this was not completed prior to enrolling into this study.

Ablative Therapy is a procedure used to destroy cancer cells and tissue. In this study Stereotactic Body Radiation Therapy (SBRT) or surgery will be used to destroy prostate cancer metastases. It is not clear if ablative therapy (SBRT or surgery) to all sites of disease used in combination with standard systemic therapy can offer better results than standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis/confirmation of prostate adenocarcinoma and no evidence of small cell cancer.
* Stage IV at presentation or relapse after curative intent therapy, classification per AJCC 8th edition: M1 disease with ≤ 5 metastases
* ≤ 3 metastases in any non-bone organ system
* Zoladex must commence within 12 weeks prior to randomization or within 12 weeks after randomization.
* Radiology (CT/MRI chest/abdomen/pelvis) within 42 days of randomization
* Bone scan within 42 days of randomization
* All tumours (Primary prostate and metastases) must be amenable to local ablative therapy (radiation and/or surgery).
* Age ≥ 18
* ECOG performance 0-2
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and economics questionnaires in either English or French
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Patients must be medically suitable for study treatments as assessed by the appropriate specialties: medical, radiation, and surgical
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* In accordance with CCTG policy, ablative therapy to metastases is to begin within 6 weeks after patient randomization
* Men of childbearing potential must have agreed to use a highly effective contraceptive method to prevent pregnancy while on study
* Patient must consent to provision of, and Investigator must confirm location of and commit to obtain a representative formalin fixed paraffin block of tumour tissue in order that the specific correlative studies described in the protocol may be conducted. Where tissue exists but local centre regulations prohibit submission of blocks of tumour tissue, the approval of the CCTG must be sought prior to randomization of the first patient to allow cores (two 2 mm cores of tumour from the block) and slides (20 x 5 micron thick unstained slides) of representative tumour tissue to be substituted
* Patient must consent to provision of samples of whole blood (for cfDNA) in order that the specific correlative studies described in the protocol may be conducted.

Exclusion Criteria:

* Prior treatment with ADT in the neoadjuvant or adjuvant setting, unless treatment was discontinued ≥ 12 months prior to randomization AND total duration of treatment was ≤ 36 months (including expiry of last depot injection).
* Previously diagnosed recurrent/metastatic disease which has been already treated with any systemic therapy or radiotherapy with palliative intent.
* Castration resistant prostate cancer, defined as rising PSA (per PCWG3) or radiographic progression in the setting of castrate levels of serum testosterone (< 1.7 nmol/L).
* Patients who present with de novo stage IV disease with pelvic lymphadenopathy as their only site of metastases (N1 M0), where the primary prostate has never been treated with curative intent prostate surgery or radiotherapy in the past.
* Inability to treat all sites of disease with local ablative therapy
* Patients with parenchymal brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 409 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-07-30 (Estimated)

PRIMARY OUTCOMES:
Failure-free Survival | 12 years
  defined as the time from randomization to the time of the first occurrence.

SECONDARY OUTCOMES:
Radiographic Progression-free Survival | 12 years
  the comparison of these outcomes between the two treatment arms will be tested by the log-rank test
Incidence of new metastases as first event | 12 years
  the comparison of these outcomes between the two treatment arms will be tested by the log-rank test
Overall Survival | 12 years
  the comparison of these outcomes between the two treatment arms will be tested by the log-rank test
Ablative treatment related adverse events (>/= grade 3) using CTCAE v5.0 | 12 years
Quality of Life measured by EORTC QLQ-C30 | 12 years
  It consists of both multi-item scales and single item measures, including five functioning domains, a global quality of life domain, three symptom domains and six single items. For each domain or single item measure a linear transformation will be applied to standardize the raw score to range between 0 and 100
Quality of Life measured by Bone Metastases module (BM22) | 12 years
  The BM22 has 22 questions consisting of the 4 subscales (painful sites (PS) and pain characteristics (PC) on the symptom scale and functional interference (FI) and psychosocial aspects (PA) on the functional scale). Modules, relevant subscales will also be linear transformed to standardize the raw score to range between 0 and 100 in accordance with the EORTC scoring manuals.
Quality of Life measured by prostate (PR25) questionnaire module | 6 years
  has 25 questions in four domains (urinary, bowel, sexual, and hormonal). Modules, relevant subscales will also be linear transformed to standardize the raw score to range between 0 and 100 in accordance with the EORTC scoring manuals.
Economic analysis measured by EQ-5D-5L | 12 years
  The robustness of the model results will be assessed using one-way and multi-way sensitivity analyses. Major drivers of medical care costs, namely hospitalization, chemotherapy and survival, will be varied ± 20%, to examine the impact on the base-case incremental cost effectiveness ratios (ICERs). Bootstrapping and the development of a cost-effectiveness acceptability curve will also be conducted.
Economic analysis by determining an incremental cost-effectiveness ratio reported as a difference in cost per FFS-year between the 2 arms | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick CF Cheung, Study Chair — Odette Cancer Centre, Sunnybrook Health Science Centre, Toronto, ON Canada; M. Tamim Niazi, Study Chair — The Jewish General Hospital, Montreal, QC Canada
Locations (18):
- Canada (18):
  - BCCA - Victoria, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
As per CCTG policy
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf